CLINICAL TRIAL: NCT03154606
Title: The Effects of Protein Source on Appetite Control, Satiety, and Subsequent Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Heather Leidy, Associate Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1701018659
Record Dates: First submitted 2017-04-19; First posted 2017-05-16 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior | interventions — calcium caseinate; Caseins; Soybean Proteins; Pea Proteins

STUDY DESIGN:
Intervention Model Description: tightly-controlled, randomized cross-over design
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HP-Beverage Breakfast (Experimental): The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will vary in protein source. All ingredients are GRAS listed and approved. All participants will complete all 12 interventions.
  Interventions: Other: Micellar Casein (#1); Other: Micellar Casein (#2); Other: Calcium Caseinate; Other: Sodium Caseinate; Other: Milk Protein Isolate; Other: Pure Protein Blend; Other: Whey Protein Isolate; Other: Native Whey Protein Isolate; Other: Soy Protein; Other: Pea Protein; Other: Native Whey: Micellar Casein (50:50) blend
- Carbohydrate Control (Active Comparator): The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will primarily as carbohydrates as a control. All ingredients are GRAS listed and approved. All participants will complete all 12 interventions.
  Interventions: Other: Carbohydrate Control

INTERVENTIONS:
Other: Micellar Casein (#1) — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from micellar casein. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Micellar Casein (#2) — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from micellar casein. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Calcium Caseinate — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from calcium casein. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Sodium Caseinate — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from sodium caseinate. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Milk Protein Isolate — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from milk protein caseinate. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Pure Protein Blend — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from pure protein blend. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Whey Protein Isolate — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from whey protein blend. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Native Whey Protein Isolate — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from Native Whey Protein Isolate. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Soy Protein — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from soy protein. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Pea Protein — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from pea protein. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Native Whey: Micellar Casein (50:50) blend — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain protein sourced predominantly from native whey: micellar casein (50:50) blend. All ingredients are GRAS listed and approved.
  Arms: HP-Beverage Breakfast
Other: Carbohydrate Control — The study participants will be provided with breakfast meals to consume. The energy content of the breakfast meals will be standardized to ~250 kcal. The meals will include the same fat content but will contain predominantly carbohydrates as a control. All ingredients are GRAS listed and approved.
  Arms: Carbohydrate Control

SUMMARY:
The investigators propose a randomized, tightly-controlled breakfast trial in normal to overweight adults that will test whether the consumption of various types of protein-rich meals, containing ~24g of protein, will differentially alter food intake and meal initiation through proposed appetite and satiety mechanisms.

Aim 1: To examine whether the consumption of protein-rich meals that vary in protein quality (source) effect:

1. postprandial feelings of hunger, fullness, desire to eat, prospective food consumption
2. postprandial fluctuations in key appetite and satiety hormones
3. eating initiation (i.e., motivation to eat (again))
4. food cravings

Aim 2: To examine whether the consumption of protein-rich meals that vary in protein quality (source) effect:

1. energy intake and food choice within the breakfast meal
2. energy intake and food choice at the next eating occasion
3. energy intake and food choice across the entire day

DETAILED DESCRIPTION:
Experimental Design: For 3 consecutive days/pattern, the participants will consume the respective treatment, at home, between 7-9 am and refrain from eating or drinking anything other than water until 12:00pm. On day 3, the participants will consume a standardized dinner at home the night before testing. On day 4, the participants will report to the research facility between 6-8 am to complete each 5-h testing day. Upon arrival to the facility, each participant will become familiarized with the testing day procedures. At time -15 min, a baseline set of computerized questionnaires (and/or blood samples) will be completed. At time +0 min, the respective breakfast treatment will be provided. Immediately following the first swallow of the breakfast meal, the participants will be given a questionnaire assessing the palatability. The participants will consume the breakfast within 20 min. After breakfast, the participants will continue to complete the questionnaires (and/or blood samples) every 30 min throughout the 5-h postprandial period. Throughout the day, the participants will also indicate if/when they would like to eat again. Regardless of the participants' meal timing request, at +240min post-breakfast, the participants will be provided with an ad libitum lunch. For the lunch meal, the participants will be given 30 min to "consume as much or as little as possible until comfortably full." Following these procedures, the participants will be allowed to leave the facility. The next day, a dietary recall will be performed to assess daily energy intake across the previous day. Lastly, on day 5 (at home), the participants will be provided with their respective breakfast along with additional carbohydrate and/or fat foods. Once the treatment breakfast is consumed, the participants can select and consume as much of the additional foods as they wish to consume within the breakfast time period (30 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* All ethnicities
* Age: 20-40y
* BMI/BMI Percentile: 18.5-29.9 kg/m2
* Consumes breakfast (>110 kcal prior to 10 am) at least 5 days/week for the past year
* Never smoked or used other tobacco products
* Willing to consume the study breakfasts
* Generally healthy (as assessed by Medical History Questionnaire)
* Health conscious as determined by answering yes to 3 pre-screening health & lifestyle questions
* Rating of ≥ 5 illustrating a minimum of "neither like nor dislike on a hedonic 9 pt taste test of all testing treatments

Exclusion Criteria:

* Clinically diagnosed with an eating disorder
* Metabolic, hormonal, and/or neural conditions/diseases that influence metabolism or appetite
* Currently or previously on a weight loss or other special diet (in the past 6 months)
* Gained/lost ≥4.5kg over the past 6 months
* Donated (or plan to donate) blood through the American Red Cross within the past 6 months (or future 6 months)
* Taking medication that would directly influence appetite (weight-loss drugs or antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months)
* Not willing or able to complete all study testing procedures
* Clinically diagnosed with a sleeping disorder

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Appetite Sensations of Hunger | 12 testing days across ~6 months
  Questionnaires assessing the appetitive sensations of hunger will be completed at specific times throughout each of the the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Appetite Sensations of Fullness | 12 testing days across ~6 months
  Questionnaires assessing the appetitive sensations of fullness will be completed at specific times throughout each of the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Appetite Sensations of Desire to Eat | 12 testing days across ~6 months
  Questionnaires assessing the appetitive sensations of desire to eat will be completed at specific times throughout each of the the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Appetite Sensations of Prospective Food Consumption | 12 testing days across ~6 months
  Questionnaires assessing the appetitive sensations of prospective food consumption will be completed at specific times throughout each of the the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.

SECONDARY OUTCOMES:
Perceived Food Cravings: Sweet | 12 testing days across ~6 months
  Questionnaires assessing the food cravings will be completed at specific times throughout each of the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Perceived Food Cravings: Salty | 12 testing days across ~6 months
  Questionnaires assessing the food cravings will be completed at specific times throughout each of the the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Perceived Food Cravings: Savory-fat | 12 testing days across ~6 months
  Questionnaires assessing the food cravings will be completed at specific times throughout each of the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Perceived Food Cravings: Meat | 12 testing days across ~6 months
  Questionnaires assessing the food cravings will be completed at specific times throughout the each of the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Perceived Breakfast Palatability | 12 testing days across ~6 months
  Questionnaires assessing the breakfast palatability will be completed at specific times throughout each of the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Perceived Energy: Sleepiness | 12 testing days across ~6 months
  Questionnaires assessing perceived sleepiness will be completed at specific times throughout each of the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Perceived Energy: Energy | 12 testing days across ~6 months
  Questionnaires assessing perceived energy will be completed at specific times throughout each of the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Perceived Energy: Alertness | 12 testing days across ~6 months
  Questionnaires assessing perceived alertness will be completed at specific times throughout each of the 4-h testing days. The questionnaires contain VAS incorporating a horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." A summation (area under the curve) will be calculated.
Food Cravings Inventory | 12 testing days across ~6 months
  Participants will fill out a Food Cravings Inventory (FCI) at 4-h post-breakfast on each testing day. The FCI is a reliable and valid self-report measure of general and specific food cravings including cravings for high fat foods, carbohydrates/starches, sweets, and fast food. The FCI defines a craving as an intense desire to consume a particular food (or food type) that is difficult to resist.
Hormonal Response to Interventions: Plasma Ghrelin | 12 testing days across ~6 months
  Ten blood samples (4 ml/sample) will be collected throughout each of the the 4-h testing days. The samples will be collected in EDTA test tubes containing pefabloc SC and DPP-IV to reduce protein degradation. Within 10-min of collection, the samples will be centrifuged, and the plasma will be stored at -80°C for future analysis.
Hormonal Response to Interventions: Plasma PYY | 12 testing days across ~6 months
  Ten blood samples (4 ml/sample) will be collected throughout each of the 4-h testing days. The samples will be collected in EDTA test tubes containing pefabloc SC and DPP-IV to reduce protein degradation. Within 10-min of collection, the samples will be centrifuged, and the plasma will be stored at -80°C for future analysis.
Hormonal Response to Interventions: Plasma GLP-1 | 12 testing days across ~6 months
  Ten blood samples (4 ml/sample) will be collected throughout each of the the 4-h testing days. The samples will be collected in EDTA test tubes containing pefabloc SC and DPP-IV to reduce protein degradation. Within 10-min of collection, the samples will be centrifuged, and the plasma will be stored at -80°C for future analysis.
24-h Energy Intake Dietary Recalls | 12 testing days across ~6 months
  To assess the participant's total energy content, macronutrient content, macronutrient consumption, and meal patterning, all subjects will complete a dietary recall following each testing day. The study staff will contact the participant the day after each of the testing days and ask questions related to the quantity, type, brand, preparation, and timing of food consumed following the testing day. Total energy content and macronutrient composition will be calculated using nutrition software.
Ad Libitum Breakfast | 12 testing days across ~6 months
  Free-living energy intake at breakfast will be assessed on day 5, of each testing period, through a meal-specific food packout . The participants will first consume the respective breakfast treatment. Additionally, the participants will be provided with an excess of macronutrient-specific foods to consume, ad libitum for the breakfast time period (30 minutes), after the required, respective breakfast treatment. All food items will be initially weighed and recorded. The participants will be instructed to return all uneaten foods as well as all wrappers and containers from consumed food. Any partially eaten, returned items will be weighed accordingly. Breakfast meal energy and macronutrient content will be assessed from these packouts.

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Leidy, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Griffith CA, Leidy HJ, Gwin JA. Indices of Sleep Health Are Associated With Timing and Duration of Eating in Young Adults. J Acad Nutr Diet. 2024 Aug;124(8):1051-1057. doi: 10.1016/j.jand.2024.04.016. Epub 2024 Apr 30. PMID 38697355
- [Derived] Braden ML, Gwin JA, Leidy HJ. Protein Source Influences Acute Appetite and Satiety but Not Subsequent Food Intake in Healthy Adults. J Nutr. 2023 Jun;153(6):1825-1833. doi: 10.1016/j.tjnut.2023.04.001. Epub 2023 Apr 6. PMID 37030593
- [Derived] Douglas SM, Leidy HJ. Novel Methodological Considerations Regarding the Use of Visual Analog Scale (VAS) Appetite Questionnaires in Tightly Controlled Feeding Trials. Curr Dev Nutr. 2019 May 2;3(6):nzz061. doi: 10.1093/cdn/nzz061. eCollection 2019 Jun. PMID 31206096